CLINICAL TRIAL: NCT04153643
Title: Arthroscopic Partial Meniscectomy Registry
Brief Title: Meniscus Surgery Registry
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leslie Bisson, June A. and Eugene R. Mindell, MD Professor and Chair of Orthopaedic Surgery, State University of New York at Buffalo
Other Study IDs: STUDY00003999
Record Dates: First submitted 2019-11-01; First posted 2019-11-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Meniscus Lesion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Arthroscopic Partial Meniscectomy — Surgical treatment for meniscus tear

SUMMARY:
The purpose of this study is to create a data registry of arthroscopic partial meniscectomies performed at our institution. This information will then be used to examine trends over time, predictive factors, and outcomes of arthroscopic partial meniscectomy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo arthroscopic partial meniscectomy with one of the study investigators at University at Buffalo Medical Doctors Orthopaedics and Sports Medicine

Exclusion Criteria:

* Non-english speaking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing arthroscopic partial meniscectomy
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Knee Pain Score | 20 years
  minimum of 0 (poor function), maximum of 100 (excellent function)

CONTACTS AND LOCATIONS:
Locations (1):
- UBMD Orthopaedics & Sports Medicine, Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: No